CLINICAL TRIAL: NCT00207610
Title: Phase 3 Study of the Prevention of Postpartum Anemia by Three Different Strategies
Brief Title: Iron Supplementation Among Low-Income Postpartum Women
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Centers for Disease Control and Prevention (U.S. Federal Agency)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: CDC-NCCDPHP-TS-0780
Record Dates: First submitted 2005-09-16; First posted 2005-09-21 (Estimated); Last update posted 2009-02-03 (Estimated); Status verified 2009-01

CONDITIONS: Anemia
Keywords: Anemia; Postpartum; iron; supplements
MeSH Terms: conditions — Anemia | interventions — Therapeutics

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

INTERVENTIONS:
Behavioral: Daily iron supplements of 65 mg a day for 3 months
Behavioral: Universal anemia screening and treatment
Behavioral: Selective anemia screening and treatment

SUMMARY:
Anemia is common among low-income women after they have given birth. Anemia, or low hemoglobin in the blood cells, is usually caused by not having enough iron. Blood cells usually carry oxygen to other parts of the body. Without enough hemoglobin, the ability of blood cells to carry oxygen is decreased. Memory and work may be impaired. The purpose of this study is to evaluate three methods of giving iron to prevent anemia among low-income women after they have given birth.

DETAILED DESCRIPTION:
Currently the Centers for Disease Control and Prevention recommendations to prevent iron deficiency advocate selective screening and treatment of anemia at about 6 weeks postpartum. However, among some groups, such as low income women, data suggest that anemia and iron deficiency are common. This study aims to evaluate the effectiveness of three stategies to prevent iron deficiency among low income postpartum women in Mississippi.

Comparisons: Clinics will be randomized to one of three strategies: 1)Selective anemia screening and treatment of anemic women, 2)universal anemia screening and treatment of anemic women, or 3)universal iron supplementation of 65 mg a day for three months.

ELIGIBILITY:
Inclusion Criteria:

* postpartum girls and women, 2-6 weeks after birth
* age 13 years or more
* WIC certified

Exclusion Criteria:

* sickle cell anemia
* Hemoglobin < 7 g/dL

Min Age: 13 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Enrollment: 959 (Actual)
Dates: Start 2003-06; Primary Completion 2007-09 (Actual); Study Completion 2007-09 (Actual)

PRIMARY OUTCOMES:
anemia | 6 months postpartum

CONTACTS AND LOCATIONS:
Overall Officials: Amal K Mitra, MD, DrPH, Principal Investigator — University of Southern Mississippi
Locations (1):
- Center for Community Health, University of Southern Mississippi, Hattiesburg, Mississippi, United States